CLINICAL TRIAL: NCT02775734
Title: N-acetyl-cysteine in Clomiphene Citrate Resistant Polycystic Ovary Syndrome After Laparoscopic Ovarian Drilling: A Randomized Controlled Trial
Brief Title: NAC in CC Resistant PCOS After LOD
Acronym: NAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS1275
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; N-acetyl-cysteine; Clomiphene citrate; Clomiphene citrate resistant; Laparoscopic ovarian drilling; therapy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Acetylcysteine; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetyl-cysteine (Active Comparator): N-acetyl-cysteine + Clomiphene citrate + LOD
  Interventions: Drug: N-acetyl-cysteine; Drug: Clomiphene citrate
- NO N-acetyl-cysteine (Active Comparator): Clomiphene citrate + LOD
  Interventions: Drug: Clomiphene citrate

INTERVENTIONS:
Drug: N-acetyl-cysteine — N-acetyl-cysteine + Clomiphene citrate + Laparoscopic ovarian drilling
  Arms: N-acetyl-cysteine
Drug: Clomiphene citrate — Clomiphene citrate + Laparoscopic ovarian drilling

SUMMARY:
This prospective randomized placebo-controlled double blind clinical trial will conducted in Ain Shams University maternity Hospital including 120 women diagnosed with clomiphene citrate resistant polycystic ovary syndrome. After laparoscopic ovarian drilling, they will be randomized to either receiving 50 mg oral clomiphene citrate twice daily and oral NAC 1,200 mg/day for 5 days starting from cycle day 2 to cycle day 6 (group 1 = 60 patients) or clomiphene citrate only (group 2 = 60 patients). The primary outcome will be biochemical pregnancy rate, secondary outcomes include Clinical pregnancy rate, ovulation rate, live birth rate, number of follicles ≥ 18 mm and endometrial thickness at triggering ovulation, mid- luteal sub-endometrial blood flow indices, and incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 30 Kg/m 2.
* CC-resistant Polycystic ovary syndrome

Exclusion Criteria:

* • Patients with BMI under 25 or over 30 Kg/m 2.

  * Hyper or hypothyroidism, or hyperprolactinemia.
  * Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs.
  * Intention to start a diet or a specific program of physical activity.
  * Organic pelvic diseases.
  * Tubal or male factor infertility.
  * Interval of earlier treatment with any of the fertility drugs of less than 6 months.
  * Contraindication to either:

    * Clomiphene citrate: liver disease, undiagnosed abnormal uterine bleeding, uterine fibroids, endometrial cancer, ovarian enlargement or hyper stimulation
    * HCG injection: ovarian enlargement or hyper stimulation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Biochemical pregnancy rate | 6 months

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 months
Live-birth rate | 15 months
Ovulation rate | 6 months
follicles more than or equal 18 mm | 6 months
Pre-ovulatory endometrial thickness | 6 months
mid-luteal sub-endometrial doppler blood flow indices | 6 months
Incidence of side effects | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided